CLINICAL TRIAL: NCT02975219
Title: Determine the Feasibility of Detecting Endometriosis During Surgery Using a Molecular Targeted Fluorescent Imaging Tracer
Brief Title: Feasibility Study of Using Molecular Fluorescence Guided Surgery in Endometriosis
Acronym: Endo-light
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, G.M. van Dam, prof. dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/304
Record Dates: First submitted 2016-11-17; First posted 2016-11-29 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): 4.5mg Bevacizumab-800CW intravenously
  Interventions: Drug: Bevacizumab-800CW

INTERVENTIONS:
Drug: Bevacizumab-800CW — 4.5mg Bevacizumab-800CW will be administered intravenously three days prior to surgery
  Other Names: Bevacizumab-IRDye800CW

SUMMARY:
Incomplete resection of endometriosis lesions often results in recurrence of symptoms and the need for repeated surgery, with considerable associated morbidity. The aim of this pilot project is to determine the feasibility of fluorescence imaging to improve the treatment of endometriosis in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged ≥ 18 years
2. Scheduled for surgery for the treatment of endometriosis
3. WHO performance score of 0-2
4. Written informed consent

   For female subjects who are of childbearing potential, are premenopausal with intact reproductive organs or are less than 2 years post-menopausal:
5. A negative serum pregnancy test prior to receiving the tracer
6. Willing to ensure that she or her partner uses effective contraception during the trial and for 6 months thereafter.

Exclusion Criteria:

1. Medical or psychiatric conditions that compromise the patient's ability to give informed consent
2. Pregnancy
3. History of infusion reactions to Bevacizumab or other monoclonal antibody therapies
4. Significant renal, cardiac, or pulmonary disease (ASA III-IV)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Tracer accumulation of bevacizumab-800cw in endometriosis lesions assessed by ex vivo measurement of the mean fluorescent intensity correlated to histopathology | within 6 months after surgery

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | within two weeks after tracer injection

CONTACTS AND LOCATIONS:
Overall Officials: Gooitzen van Dam, prof dr, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands